CLINICAL TRIAL: NCT04420403
Title: Investigation of the Effectiveness of Manual Therapy Plus Cervical Stabilization Exercise on Balance, Proprioception, and Neck Muscle Morphology in Chronic Neck Pain
Brief Title: Investigation of the Effectiveness of Manual Therapy Plus Cervical Stabilization Exercise in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, associate professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/05/28
Record Dates: First submitted 2020-05-29; First posted 2020-06-09 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Neck Pain
Keywords: neck pain; manual therapy; exercise; postural control
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to manual therapy plus cervical stabilization exercise group (intervention group) and only the manual therapy group (control group).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy plus cervical stabilization exercise group (Experimental): The patients diagnosed with chronic neck pain (CNP) with 18-55 years of age followed by routine controls and who were volunteered will be included in the study.
  Interventions: Other: Manual Therapy; Other: Cervical Stabilazation Exercise (CSE)
- Only manual therapy group (Active Comparator): The patients diagnosed with CNP with 18-55 years of age followed by routine controls and who were volunteered will be included in the study.
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Manual Therapy — Cyriax's mobilization techniques will be applied as manual therapy. Before the mobilization, soft tissue mobilization techniques will be applied to relieve muscular spasm and preventing the patient' s anxiety. Bringing, manual traction, manual traction with rotation, manual traction with anterior-posterior gliding and lateral gliding mobilization techniques will be applied. Appropriate mobility techniques will be selected according to the complaints and symptoms of the patients. Cervical mobilization applications will take an average of 15-20 minutes.
Other: Cervical Stabilazation Exercise (CSE) — The CSE program aims to maintain a neutral spine position and activate deep cervical muscles during exercises. It is performed in stages with gradual progression according to the stages of motor learning and sensory-motor integration, namely, static, dynamic, and functional. The program will start with postural training and then the cervical bracing technique with the activation of deep neck flexors for CSE was performed. The patients will be asked to maintain a neutral spine during the exercises and throughout the day as much as possible. The difficulty and variety of exercises will be increased weekly. It will be carried out 2 days a week for 6 weeks (12 sessions) by the supervisor physiotherapist.
  Arms: Manual therapy plus cervical stabilization exercise group

SUMMARY:
This study aims to investigate the effectiveness of manual therapy plus cervical stabilization exercise compared to manual therapy alone on balance, proprioception, and neck muscle morphology in chronic neck pain.

DETAILED DESCRIPTION:
Neck pain is defined as pain and/or stiffness localized to the dorsal area of the area between the condyle of the occiput and the third thoracic vertebra. Chronic neck pain (CNP), defined as persistent pain lasting three or more mounts, causes disability and a reduction in life quality. Balance disorders or postural instability, a deficit in proprioception, changes in muscle recruitment, a decrease in dimension of deep cervical muscle, and an increase in stiffness of superficial neck muscle may lead to pain in patients with CNP. Both manual therapy and exercise have favorable effects on management with CNP. According to our knowledge, no study has investigated the effects of manual therapy plus cervical stabilization exercise on balance, proprioception, and neck muscle morphology in CNP, yet.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 55 years of age,
* Having generalized neck pain for more than 3 months,
* Being volunteer

Exclusion Criteria:

* Being pregnant,
* Malignancy,
* Having cervical stenosis,
* Severe cervical spondylosis,
* Cervical fractures and tumor,
* Osteoporosis,
* Positive vertebrobasilar test
* Positive Babinski reflex
* Neurologic deficit related to compression of the spinal root or cord,
* Having neurologic, dermatologic, infectious, inflammatory rheumatologic and endocrine diseases,
* Being an inability to fulfill the questionnaires,
* Any problems that will hinder exercise (advanced cardiopulmonary or orthopedic problems), having intervention including exercise program or physiotherapy in the three months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Balance | change from baseline at 6 weeks
  The balance will be evaluated with Biodex BioSwayTM Balance Evaluation System. It reliably measures the patient's ability to balance on soft and/or hard ground.

SECONDARY OUTCOMES:
Proprioception | change from baseline at 6 weeks
  Proprioception will be assessed with dual digital inclinometer. The feet of the inclinometers will be placed as simultaneously as possible over the head of the patients and the cervical seventh vertebra. Firstly, patients will be asked to move their heads forward as possible as from the neutral position and then they will try to find neutral position from reached position. The angle on digital display of inclinometer will be recorded as degree. Each test will be repeated 3 times and the average deviation error score will be recorded.
Muscle morphology | change from baseline at 6 weeks
  The thickness and stiffness of the neck muscles will be evaluated by a specialist radiologist with real-time ultrasonography. It is a reliable, valid and, non-invasive method that provides an assessment of muscle morphology. Measurements will be made by using the Logiq S7 / Expert ultrasound device. The cross-sectional area of deep neck muscle with sonography, the stiffness of the superficial muscles with elastography were assessed.
Pain intensity | change from baseline at 6 weeks
  The pain intensity will be assessed with the Visual Analog Scale, which consists of a horizontal line of 10 cm in length. For pain level assessment, "0" defines "no pain" and "10" defines "unbearable pain''. The participants will be asked to mark the intensity of their pain level.
Disability level | change from baseline at 6 weeks
  The disability level will be measured with the Turkish version of Neck Disability Index (NDI). It consists of 10 sections which include the severity of pain, personal care, lifting, reading, headache, concentration, work-life, driving, sleeping and leisure activities. There are 6 responses for each section, scored 0 (no pain and no functional limitation) and 5 (worst pain and maximum limitation). The total score ranges from 0 to 50. Patients will be asked to select the most appropriate option for each section.

CONTACTS AND LOCATIONS:
Overall Officials: seyda toprak celenay, PhD, PT, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No